CLINICAL TRIAL: NCT04028648
Title: Generation of Prediction Equations to Analyze Body Composition of the Elderly Based on Bioelectrical Impedance Analysis (BIA)
Brief Title: Generation of Prediction Equations for BIA of the Elderly
Status: Completed | Type: Observational
Sponsor: Seca GmbH & Co. Kg. (Industry)
Responsible Party: Sponsor
Other Study IDs: BCA-12
Record Dates: First submitted 2018-09-14; First posted 2019-07-22 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-10

CONDITIONS: Healthy Elderly

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- elderly: 150 elderlies (>60 years): community dwelling or living in old

SUMMARY:
The objective of the study is to develop prediction equations for calculating Fat-Free Mass FFM, Total Body Water TBW, Extracellular Water ECW, Visceral Adipose Tissue VAT, total Skeletal Muscle Mass SMM and segmental SMM in a group of elderly. The prediction equations are based on linear regression analysis between the gold standard reference methods Air Displacement Plethysmography ADP, Dual-energy X-ray Absorptiometry DXA, Magnet Resonance Imaging MRI, Deuterium dilution method (D2O) and Sodium Bromide dilution method (NaBr) on the one hand and bioelectrical impedance measurements on the other hand.

Multi-frequency bioimpedance is measured for all body segments: right arm, left arm, right leg, left leg, trunk, right body side and left body side using the seca mBCA 515 in standing position and the seca mBCA 525 in standing and lying position.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects older than 60 years,
* stable medication (no changes during the past 6 months),
* subjects need to be able to sign the informed consent and privacy policy

Exclusion Criteria:

* acute disease
* intake of diuretics
* wearing of support stockings
* edema diagnosed by inspection and palpation of lower limbs
* paralysis e.g. after a stroke
* neurodegenerative diseases e.g. ALS
* tumors in treatment
* amputation
* electronic implants e.g. pacemaker
* under the skin applied injection systems (e.g. insulin pumps or pain pumps)
* probands who cannot provide an ICF by themselves
* probands who might be dependent from the sponsor or the investigation site
* current alcohol abuse
* active prostheses
* electronic life-support systems, e.g. artificial heart, artificial lung
* portable electronic medical devices, e.g. ECG devices or infusion pumps
* metallic implants
* cochlea implants und heart valves prothesis (e.g. Starr-Edwards-Prothesis)
* vessel clips in the brain or medulla applied before 1995
* defeatable pumps
* catheter
* iron or metallic parts in the body (e.g. shard of metal)
* dental braces
* magnetic tooth implants
* not removeable piercings
* extensive tattoos

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 150 elderlies (>60 years): community dwelling or living in old nursing homes
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Human Nutrition and Food Science, Kiel, Germany

REFERENCES:
- [Derived] Enderle J, Reljic D, Jensen B, Peine S, Zopf Y, Bosy-Westphal A. Normal values for body composition in adults are better represented by continuous reference ranges dependent on age and BMI. Clin Nutr. 2023 May;42(5):644-652. doi: 10.1016/j.clnu.2023.03.006. Epub 2023 Mar 9. PMID 36933351

RESULTS

PARTICIPANT FLOW:
Groups:
- Elderly: 150 elderlies (>60 years): community dwelling or living in old people's homes.
Period: Overall Study
Arm/Group | Elderly
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Elderly
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight [Mean (Standard Deviation); unit: kg] | 74.3 (16.3)

OUTCOME MEASURES:

1. Primary Outcome: Total Body Water
Description: Total body water (TBW) by deuterium (D2O) dilution
Time Frame: 15 minutes
Measure: Least Squares Mean (Standard Deviation); unit: liter
Arm/Group | Elderly
Number analyzed (Participants) | 150
liter | 1.85 (0.11)

2. Primary Outcome: Extracellular Water
Description: Extracellular water (ECW) by NaBr dilution
Time Frame: 15 minutes
Measure: Least Squares Mean (Standard Deviation); unit: liter
Arm/Group | Elderly
Number analyzed (Participants) | 150
liter | 0.74 (0.04)

3. Primary Outcome: Fat-free Mass
Description: Fat-free mass by a 4-compartment model based on dual energy x-ray absorption (DXA), air displacement plethysmography (ADP), D2O dilution and weight
Time Frame: 15 minutes
Measure: Least Squares Mean (Standard Deviation); unit: kg
Arm/Group | Elderly
Number analyzed (Participants) | 150
kg | 2.20 (0.13)

4. Primary Outcome: Skeletal Muscle Mass
Description: Skeletal muscle mass (SMM) by magnetic resonance imaging (MRI)
Time Frame: 1 hour
Measure: Least Squares Mean (Standard Deviation); unit: kg
Arm/Group | Elderly
Number analyzed (Participants) | 150
kg | 2.07 (0.12)

5. Primary Outcome: Visceral Adipose Tissue
Description: Visceral adipose tissue (VAT) by magnetic resonance imaging MRI
Time Frame: 1 hour
Measure: Least Squares Mean (Standard Deviation); unit: liter
Arm/Group | Elderly
Number analyzed (Participants) | 150
liter | 0.92 (0.05)

ADVERSE EVENTS:
Time Frame: 2 days (During the presence in the research facility. 1 day for all measurements except MRI, 1 day for MRI.)
Arm/Group | Elderly
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT04028648/Prot_SAP_000.pdf